CLINICAL TRIAL: NCT01106183
Title: A Double Blind Study on the Efficacy of a Colostrum and Egg Yolk Supplement vs. Placebo to Reduce Frequency and Duration of Upper Respiratory Tract Infections in Healthy Adults
Brief Title: Efficacy of Transfer Factor to Prevent Upper Respiratory Tract Infections in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 38766 4Life-Transfer Factor
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2011-11

CONDITIONS: Upper Respiratory Tract Infections Due to Influenza or Rhinovirus
MeSH Terms: interventions — Transfer Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transfer Factor (Active Comparator): Transfer factor supplement; 2 capsules per day
  Interventions: Dietary Supplement: transfer factor
- Sugar pill (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: transfer factor — capsules, 2 per day by mouth for 7 weeks.
  Arms: Transfer Factor
Dietary Supplement: Placebo — cornstarch, 2 capsules per day by mouth.
  Arms: Sugar pill

SUMMARY:
The goals of our study are to critically evaluate if a healthy population supplemented with Transfer factor experiences fewer incidences of colds and flu, or experience shorter duration of illness compared to an identical population taking placebo. In this study we will give either Transfer factor or a placebo to two groups of healthy adult men and women for a period of 7 weeks in a double-blind experimental design. The frequency and duration of colds and flu-like symptoms will be recorded during the course of the study. Saliva samples will be collected weekly and assessed for salivary IgA secretion rate. Data from this study will establish the efficacy of Transfer Factor to support a healthy immune system.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (18 - 40) who are in good health

Exclusion Criteria:

* Subjects who are allergic to eggs (on which the supplement is based). If a volunteer is not sure if they are allergic to eggs or milk. Those who are currently smoking, have cardiovascular disease, cancer, diabetes, liver disease, renal insufficiency, any chronic disease that might interfere with study participation, BMI above 40 kg/m2, consumption of >12 alcoholic drinks weekly, or unwillingness to stop current supplement intake. Women who are pregnant or lactating will also be excluded from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States